# **Protocol**

# Tenecteplase in Wake-up Ischaemic Stroke Trial (TWIST)

A randomised-controlled trial of thrombolytic treatment with tenecteplase for acute ischaemic stroke upon awakening

> EudraCT number: 2014-000096-80 Sponsor's protocol code number: 01

#### **Sponsor:**

University Hospital of North Norway, NO-9038 Tromsø, Norway Telephone number: +47 77626000

#### **Trial Coordinating Centre:**

Brain and Circulation Research Group, Department of Neurology, University Hospital of North Norway, and Faculty of Health Sciences, University of Tromsø Address: Department of Neurology, University Hospital of North Norway, NO-9038 Tromsø, Norway

Telephone number: +47 77627120

# Signature page

| Sponsor |
|---|
| Director of Research (signature and date) University Hospital of North Norway |
| Trial Coordinating Investigator and Head of Brain and Circulation Research Group (signature and date) |
| University Hospital of North Norway and University of Tromsø |
| Principal investigator |
| I have read this protocol and agree that it contains all the necessary details for carrying out the study. I will conduct the study as outlined herein and will complete the study within the time designated. |
| I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of the study. I will discuss this material with them to ensure that they are fully informed regarding the study intervention and the conduct of the study. |
| Principal investigator (signature and date) |
| Name of institution |

# 1. Contents

| 1. | Cont | tents | 3 | |
|---|---|---|---|---|
| 2. | Sum | mary | 5 | |
| 3. | Back | reground and rationale | 5 | |
| 3 | .1 | Introduction | | 5 |
| 3 | .2 | Potential benefits and harms of tenecteplase | | 5 |
| 3 | .3 | Multi-modal CT for the selection or patients to thrombolytic therapy | | |
| 4. | Trial | l design, questions, and hypotheses | | |
| | .1 | Trial design | | 8 |
| 4 | .2 | Study questions and objectives | | |
| 4 | .3 | Hypotheses | | |
| | | y population | | |
| | .1 | Inclusion criteria. | | 8 |
| | .2 | Exclusion criteria | | |
| _ | | ent screening | | , |
| | .1 | Patient screening. | | 9 |
| _ | .2 | Non-contrast CT and CT angiography for patient screening before randomisation | | |
| _ | .3 | CT perfusion at selected centres before randomisation (substudy) | | |
| | .4 | Routine use of MRI before randomisation (substady) | | |
| | | ent inclusion | | 10 |
| | .1 | Patient information and consent/assent | | 10 |
| | .2 | Randomisation procedure and recording of baseline characteristics | | |
| 8. | | I treatment | | 10 |
| ο. | 8.1 | Open-label tenecteplase plus best standard care | | 11 |
| | 8.2 | Best standard care alone | | |
| | 8.3 | Best standard care and other treatments | | |
| Λ | 8.4 | Management of serious adverse events related to study treatment | | 11 |
| 9. | | ts and examinations from trial entry till end of follow-up | | 10 |
| | 9.1 | Visits and examinations during stay in hospital | | |
| | 9.2 | Centralised follow-up via telephone or mail at 3 months (90 ±7 days) | 1 | 12 |
| 1.0 | 9.3 | Long-term follow-up by record linkage with central registries | | 22 |
| | | ct variables | | 1.2 |
| | 0.1 | Primary effect variable | | |
| | 0.2 | Secondary effect variables | | 13 |
| | | lysis and statistical considerations | | |
| | 1.1 | 1 | | |
| | 1.2 | | 1.5 | 14 |
| | | l conduct and practices/procedures | | |
| | 2.1 | Compliance with regulations and guidelines | | |
| | 2.2 | Data protection | | |
| | 2.3 | Ethical conduct | | |
| | 2.4 | Liability | | |
| | 2.5 | Recording and reporting of serious adverse events | | |
| | 2.6 | Event adjudication | | |
| | 2.7 | Monitoring of data quality | | |
| | 2.8 | Handling of protocol violations and protocol amendments | | |
| | 2.9 | Monitoring of effectiveness and safety | | |
| 1 | 2.10 | Audit and inspection. | | |
| | 2.11 | Handling of patient data | | |
| | 2.12 | Handling of the list of treatment codes | | |
| | 2.13 | Screening logs | | |
| | | Financial conduct. | | |
| | | Publication and data sharing policy | | |
| | | User involvement | | 17 |
| 13. | Cent | ral trial organisation | | |
| 1 | 3.1 | Sponsors and funding bodies | | 17 |

| 13.2 | Trial Coordinating Centre | 18 |
|---|---|---|
| 13.3 | Trial Statistical Centre | 18 |
| 13.4 | Executive Committee | 18 |
| 13.5 | Imaging Scientific Committee | 18 |
| 13.6 | Trial Steering Committee | |
| 13.7 | Data Monitoring Committee | 18 |
| 13.8 | Event Adjudication Committee | 18 |
| 14. Tim | e table and end of trial | 18 |
| 15. Refe | erences | 19 |
| 16. App | endix | 23 |
| 16.1 | On-going studies of thrombolytic treatment for wake-up stroke | 23 |
| 16.2 | Definitions of clinical events | 23 |
| 16.2 | | |
| 16.2 | .2 Death | 23 |
| 16.2 | Recurrent stroke | 24 |
| 16.2 | 2.4 Symptomatic intracranial haemorrhage | 24 |
| 16.2 | 2.5 Asymptomatic intracranial haemorrhage | 24 |
| 16.2 | · · | |
| 16.2 | | |
| 16.2 | | |
| 16.3 | Abbreviations | |
| 17. Sum | nmary of changes | 25 |
| 17.1 | Protocol version/date 160323 | |
| 17.2 | Protocol version/date 160421 | 26 |
| 17.3 | Protocol version/date 170412 | 26 |
| 17.4 | Protocol version/date 180410 | 26 |
| 17.5 | Protocol version/date 180704 | 26 |
| 17.6 | Protocol version/date 200131 | 26 |
| 17.7 | Protocol version/date 200917 | 26 |

# 2. Summary

Tenecteplase in Wake-up Ischaemic Stroke Trial (TWIST) is a randomised-controlled, open-label trial of thrombolytic treatment with tenecteplase for acute ischaemic stroke upon awakening.

The trial aims to answer the following questions:

- Can thrombolytic treatment with tenecteplase given within 4.5 hours of wake-up reduce the risk of poor functional outcome at 3 months?
- Can findings on non-contrast CT and CT angiography (and CT perfusion at selected centres) identify patients who benefit from such treatment, compared to patients without such findings?

Patients are eligible if they have ischaemic stroke causing measurable neurologic deficits, and can be given tenecteplase within 4.5 hours after awakening. Patients will undergo brain CT and CT angiography (if possible) to exclude large infarction or other contraindications to thrombolytic treatment. Non-contrast CT and CT angiography (if possible) will be repeated on day 2.

Patients will be allocated to tenecteplase 0.25 mg/kg as a bolus (maximum dose 25 mg) or to control. The primary effect variable is functional outcome at 3 months, as measured by the modified Rankin Scale (mRS).

The target is to include a total of 600 patients from centres in Norway, Sweden, Denmark, Finland, Estonia, Lithuania, Latvia, Switzerland, New Zealand and the United Kingdom. The sponsor of the trial is University Hospital of North Norway.

# 3. Background and rationale

#### 3.1 Introduction

Thrombolytic treatment with recombinant tissue plasminogen activator (rt-PA) given within 4.5 hours of onset improves clinical outcome after ischaemic stroke, despite an increased risk of intracranial haemorrhage.<sup>1,2</sup> Patients who have new stroke symptoms when they wake up from sleep ("wake-up stroke") are excluded for such treatment, because the time of stroke onset is unknown. About one in five strokes occur during sleep,<sup>3-5</sup> and it is unknown whether patients with wake-up stroke will benefit from thrombolytic treatment.

There are reasons to expect that patients with wake-up stroke will benefit from treatment. Several studies have shown that the onset of stroke during sleep is close to awakening, <sup>6,7</sup> and that patients with wake-up stroke share many clinical and radiological findings with patients with stroke duration less than 4.5 hours. <sup>8-13</sup> Studies have also shown that thrombolytic treatment is safe in patients with wake-up stroke up to 4.5 hours from wakening, <sup>14-19</sup> and recently the WAKE-UP trial showed benefit of treatment with alteplase in patients selected based on DWI/FLAIR mismatch on MRI. <sup>20</sup> In a Cochrane systematic review<sup>21</sup> we have identified only one completed, small randomised-controlled trial of only nine patients. <sup>22</sup> Two trials have recently been completed (EXTEND, <sup>23</sup> THAWS, <sup>24</sup>) and one is on-going (WASSABI, <sup>25</sup> see Appendix). All these three trials use alteplase, and all use advanced imaging techniques for selection of patients. We will use a different strategy, and perform a large trial of tenecteplase, using a pragmatic study design, without exclusion of patients based on MRI findings. The trial will be complementary to the other trials, and is planned in advance to be included in our Cochrane meta-analysis of all trials of thrombolytic treatment for wake-up stroke, so that smaller, but still worthwhile effects can be detected that may be missed by the individual trials.

#### 3.2 Potential benefits and harms of tenecteplase

Pharmacological properties

Tenecteplase is an alteplase molecule that is genetically engineered to have pharmacological advantages over alteplase: it has a 14-fold greater fibrin specificity and a very rapid onset of action compared to alteplase, has a longer half-life, and can be given as a single bolus, whereas alteplase must be given as a continuous infusion over one hour. Tenecteplase also has a smaller effect on plasma fibrinogen levels, which is beneficial for avoidance of intracranial haemorrhage, and weaker pro-thrombotic effects. Which is defected as a smaller effect of the same pro-thrombotic effects.

#### Data from pre-clinical studies

Animal models have shown that tenecteplase acts faster<sup>33</sup> and more potent<sup>33-35</sup> than alteplase, and that tenecteplase produces a more rapid and complete recanalisation of occluded arteries. <sup>31,34,36</sup> Models have also shown that experimentally induced infarcts were less frequently converted to haemorrhage with tenecteplase than with bio-equivalent doses of alteplase<sup>36,37</sup> and that the risk peripheral or major haemorrhage<sup>31</sup> and intracranial haemorrhage<sup>36-41</sup> was equal to or lower than the risk with alteplase.

#### Data from clinical studies

Tenecteplase is preferred over alteplase for treatment of myocardial infarction, because it has lower risk of bleeding complications, and because of the pharmacological advantages listed above.<sup>42</sup>

A number of observational studies in patients with ischaemic stroke have shown that, compared to alteplase, tenecteplase is associated with similar or better recanalisation rates and clinical outcomes, and a similar or lower risk of intracranial haemorrhage. A3-47 These studies have also concluded that the optimal dose of tenecteplase for stroke is 0.25 mg/kg. 28,45,48,49

There has also been three small randomised-controlled trials of tenecteplase vs. alteplase in acute ischaemic stroke. 45,47,48 Meta-analysis of these trials with a total of 283 patients have shown that 76/178 patients (43%) patients given tenecteplase (doses ranging from 0.1 to 0.4 mg/kg) achieved good functional outcome (mRS score 0-1), compared to 33/105 patients (31%) patients given alteplase (odds ratio (OR) 1.39, 95% confidence interval (CI) 0.82-2.36, Figure 1).

Figure 1. Good functional outcome (mRS score 0-1) at three months

| | Tenecteplase (any | dose) | Altepl | ase | | Odds Ratio | Odds Ratio |
|---|---|---|---|---|---|---|---|
| Study or Subgroup | Events | Total | Events | Total | Weight | M-H, Random, 95% CI | M-H, Random, 95% CI |
| ATTEST 2014 | 13 | 47 | 10 | 49 | 31.2% | 1.49 [0.58, 3.83] | |
| Clarke Haley 2010 | 36 | 81 | 13 | 31 | 39.6% | 1.11 [0.48, 2.56] | <del></del> |
| Parsons 2012 | 27 | 50 | 10 | 25 | 29.2% | 1.76 [0.66, 4.67] | +- |
| Total (95% CI) | | 178 | | 105 | 100.0% | 1.39 [0.82, 2.36] | • |
| Total events | 76 | | 33 | | | | |
| Heterogeneity: Tau2 = | : 0.00; Chi <sup>2</sup> = 0.53, d | df = 2 (F | P = 0.77 | $I^{2} = 0$ | % | | 0.01 0.1 1 10 100 |
| Test for overall effect: | Z = 1.23 (P = 0.22) | | | | | | Favours Alteplase Favours Tenecteplase |

There was also a non-significant lower risk of symptomatic intracranial haemorrhage in patients given tenecteplase (Figure 2). The risks were 7/131 (5%) in patients given tenecteplase and 4/56 (7%) in patients given alteplase (OR 0.71, 95% CI 0.11-4.42). ATTEST 2014 did not provide data on symptomatic intracranial haemorrhage.

Figure 2. Symptomatic intracranial haemorrhage



There was no significant difference in the risk of death at three months (Figure 3). In total, 24 of the 178 patients (13%) given tenecteplase and 17 of the 123 patients (14%) given alteplase were dead at three months (OR 1.00, 95% CI 0.52-1.95).

Figure 3. Death of all causes at three months



Another meta-analysis comparing different doses of tenecteplase concluded that 0.25 mg/kg is the preferred dose over alteplase. <sup>50</sup> There are also observational studies that support this conclusion. <sup>28,49</sup> Furthermore, an analysis of pooled data for tenecteplase 0.25 mg/kg compared to alteplase 0.9 mg/kg showed trends in favour of tenecteplase. <sup>50</sup> Tenecteplase had higher odds than alteplase for neurological improvement at 24 hours (OR 3.3, 95% CI 1.5-7.2, p=0.09), excellent clinical outcomes at three months (OR 1.9, 95% CI 0.8-4.4, p=0.3), and good clinical outcomes at three months (OR 1.9, 95% CI 0.5-7.2, p=0.4); also, tenecteplase had a lower risk of brain haemorrhage than alteplase (OR 0.3, 95% CI 0.2-1.8, p=0.4). Recently, NOR-TEST showed no difference in functional outcome at three months between patients with ischaemic stroke treated with tenecteplase 0.4 mg/kg or alteplase 0.9 mg/kg within 4.5 hours <sup>51</sup> and the EXTEND-IA TNK trial showed that tenecteplase 0.25 mg/kg was superior to alteplase 0.9 mg/kg in improving recanalisation and functional outcome at three months when given within 4.5 hours and prior to intra-arterial intervention. <sup>52</sup> Other trials of tenecteplase in patients with acute ischaemic stroke are ongoing: TASTE<sup>53</sup>, TEMPO-2<sup>54</sup> and ATTEST2. <sup>55</sup>

#### Conclusion: Potential benefits and harms of tenecteplase

The bolus administration and the very rapid onset of action makes tenecteplase an attractive option for patients with wake-up stroke, because the time to recanalisation of an occluded cerebral artery can be reduced by up to one hour, compared to alteplase. Available data from pharmacological in-vitro studies, pre-clinical studies and clinical studies also indicate that tenecteplase 0.25 mg/kg is at least as safe and at least as effective as alteplase for the treatment of acute ischaemic stroke. The favourable profile of tenecteplase seen in these studies and in studies of acute myocardial infarction, in combination with the pharmacological characteristics and advantages of bolus administration, provides a good rationale for testing tenecteplase in patients with wake-up stroke.

#### 3.3 Multi-modal CT for the selection of patients to thrombolytic therapy

The WAKE-UP trial and three other trials of thrombolytic treatment for wake-up stroke use/used advanced imaging techniques for selection of patients. <sup>20,23-25</sup> Two trials (WASSABI<sup>25</sup> and EXTEND<sup>23</sup>) use CT or MRI perfusion techniques to identify patients with ischaemic penumbra. The penumbra is an area of ischaemic, but still viable brain tissue surrounding the core of a cerebral infarction, which is assumed to be salvageable if blood flow can be promptly restored. The WAKE-UP trial<sup>20</sup> and the THAWS<sup>24</sup> used DWI/FLAIR mismatch on MRI to select patients. Infarct changes on DWI are thought to represent alterations to water diffusion and can be visualised within minutes of onset. Infarct changes on FLAIR are thought to represent cytotoxic oedema and cannot be identified until a few hours after onset. Findings suggestive of ischaemic stroke on DWI, but absence of such findings on FLAIR (DWI/FLAIR mismatch), may therefore identify patients with a short time since onset of cerebral infarction.

Demonstration of penumbra or DWI/FLAIR mismatch identifies patients with a good prognosis, but it does not necessarily identify patients with a better response to thrombolytic treatment than other patients. Only one randomised-controlled trial (MR RESCUE, of intra-arterial interventions) has examined the value of advanced imaging for patient selection<sup>56</sup>, but did not find a better effect of therapy in patients with penumbra, than in patients without penumbra.<sup>56</sup>

On the contrary, there is a risk that selection of patients based on such techniques will exclude patients from receiving an effective treatment. First, it is possible that patients without these specific radiological findings benefit equally well as those who are selected for participation in these trials, as indicated in a recent study. <sup>19</sup> Second, the techniques are far from perfect in characterising patients, for example, DWI/FLAIR mismatch can be absent in as many as 40% of patients with known stroke duration of less than three hours. <sup>57</sup> Third, these MRI techniques are time-consuming and are not available in the emergency setting in many hospitals, which means that time to thrombolytic treatment will be increased, and that some patients will be denied thrombolytic treatment altogether.

We will therefore base patient inclusion on wider and more pragmatic criteria, such as time since wake-up in combination with accepted CT exclusion criteria. Inclusion based on wider criteria will avoid excluding a large number of patients that might benefit from treatment. This will make the results applicable to patients that are encountered in everyday clinical practice, and will dramatically increase the proportion of stroke patients who can be treated. Patient can be included based on non-contrast CT alone, but CT angiography can be routinely done in many hospitals, can be done without significant delay, and can give information that will help in the selection of patients with wake-up stroke for thrombolytic treatment. <sup>58-62</sup>

# 4. Trial design, questions, and hypotheses

#### 4.1 Trial design

Randomised-controlled, open-label trial of tenecteplase in patients with acute ischaemic stroke upon awakening.

## 4.2 Study questions and objectives

The objectives of the trial is to answer the following questions, for patients who have an acute ischaemic stroke upon awakening:

- Can thrombolytic treatment with tenecteplase given within 4.5 hours of wake-up reduce the risk of poor functional outcome at 3 months?
- Can findings on non-contrast CT and CT angiography (and CT perfusion at selected centres) identify patients who benefit from such treatment, compared to patients without such findings?

#### 4.3 Hypotheses

- Thrombolytic treatment with tenecteplase will reduce the risk of poor functional outcome at 3 months. For details about size of effect, see Statistical calculations, below.
- CT angiography and CT perfusion identifies patients who benefits more from tenecteplase than other patients

# 5. Study population

Patients with acute ischaemic stroke upon awakening who can be given treatment within 4.5 hours after awakening.

#### 5.1 Inclusion criteria

- Stroke symptoms on awakening that were not present before sleep
- Clinical diagnosis of stroke with limb weakness with NIHSS score ≥3, or dysphasia
- Treatment with tenecteplase is possible within 4.5 hours of awakening
- Written consent from the patient, non-written consent from the patient (witnessed by non-participating health care personnel), or written consent from the nearest family member

#### 5.2 Exclusion criteria

- Age <18 years
- NIHSS score >25 or NIHSS consciousness score >2, or seizures during stroke onset
- Findings on non-contrast CT that indicate that the patient is unlikely to benefit from treatment:
  - Infarction comprising more than >1/3 of the middle cerebral artery territory on noncontrast CT or CT perfusion
  - Intracranial haemorrhage, structural brain lesions which can mimic stroke (e.g cerebral tumour)
- Active internal bleeding of high risk of bleeding, e.g.:
  - Major surgery, trauma or gastrointestinal or urinary tract haemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days
  - Any known defect in coagulation, e.g. current use of vitamin K antagonist with an INR >1.7 or prothrombin time >15 seconds, or use of direct thrombin inhibitors or direct factor Xa inhibitors during the last 24 hours (unless reversal of effect can be achieved by agents such as idarusizumab) or with elevated sensitive laboratory tests (such as aPTT, INR, platelet count, eucarin clotting time, TT, or appropriate factor Xa activity assays), or heparins during the last 24 hours or with an elevated aPTT greater than the upper limit of normal
  - Known defect of clotting or platelet function or platelet count below 100,000/mm<sup>3</sup> (but patients on antiplatelet agents can be included)
  - Ischaemic stroke or myocardial infarction in previous 3 months, previous intracranial haemorrhage, severe traumatic brain injury or intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm, arteriovenous malformation or aneurysm
- Contraindications to tenecteplase, e.g., acute bacterial endocarditis or pericarditis; acute pancreatitis; severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension; active hepatitis; systemic cancer with increased bleeding risk; haemostatic defect including secondary to severe hepatic, renal disease; organ biopsy; prolonged cardiopulmonary resuscitation > 2 min (within 2 weeks)
- Persistent blood pressure elevation (systolic ≥185 mmHg or diastolic ≥110 mmHg), despite blood pressure lowering treatment
- Blood glucose <2.7 or >20.0 mmol/L (use of finger-stick measurement devices is acceptable)
- Pregnancy, positive pregnancy test, childbirth during last 10 days, or breastfeeding. In any woman of childbearing potential, a pregnancy test must be performed and the result assessed before trial entry
- Other serious or life-threatening disease before the stroke: severe mental or physical disability (e.g. Mini Mental Status score  $\leq$ 20, or mRS score  $\geq$ 3), or life expectancy less than 12 months
- Patient unavailability for follow-up (e.g. no fixed address)

# 6. Patient screening

#### 6.1 Patient screening

All patients who are admitted with new stroke symptoms on awakening should be screened for inclusion into the trial. Patients will be evaluated for vital signs, physical examination, neurological status (NIHSS), ECG and CT with CT angiography (section 6.2). Routine blood tests will include blood glucose and prothrombin time/INR\*, aPTT\*, TT and/or eucarin clotting time if it is suspected the patient is taking direct thrombin inhibitors or direct factor Xa inhibitors.

<sup>\*</sup>Although it is desirable to know the results of these tests before giving intravenous tenecteplase, fibrinolytic therapy should not be delayed while awaiting the results unless (1) there is clinical suspicion of a bleeding abnormality or thrombocytopenia, (2) the patient has received heparin or warfarin within 48 hours, or (3) the patient has received other anticoagulants/direct thrombin inhibitors or direct factor Xa inhibitors.

# **6.2** Non-contrast CT and CT angiography for patient screening before randomisation

All patients should be screened with non-contrast CT, and CT angiography should be performed, if possible. Findings on non-contrast CT shall only be used to exclude patients who are unlikely to benefit from treatment (See Exclusion criteria in Section 5). If other, advanced imaging examinations are used (see sections 6.3 and 6.4, below), findings on such examinations shall not influence the decision to include the patient, unless the results of such imaging show that the patient should or should not receive thrombolytic treatment, in the opinion of the investigator.

#### 6.3 CT perfusion at selected centres before randomisation (substudy)

Some centres routinely use CT perfusion in patients with wake-up stroke, and these centres will be invited to participate in a substudy of CT perfusion. All CT scans taken in the trial will be sent to the Trial Co-ordinating Centre for central, blinded analysis.

#### 6.4 Routine use of MRI before randomisation

Some centres routinely use MRI perfusion or MRI DWI/FLAIR in patients with wake-up stroke. These examinations are not part of the trial, but MRI examinations done of patients included into the trial shall be sent to the Trial Coordinating Centre for central, blinded analysis. Extra brain scanning (CT perfusion or MRI) must not delay treatment, and we will discourage extra scanning if randomisation is delayed more than 20 minutes.

#### 7. Patient inclusion

#### 7.1 Patient information and consent/assent

Written, informed consent will be sought from all eligible patients. If the patient can consent but cannot sign, non-written consent from the patient (witnessed by non-participating health care personnel) can be accepted. If the patient is unable to consent, his/her legal representative and/or next of kin can consent on the patient's behalf depending on national legislation. The regulations governing these procedures may vary from jurisdiction to jurisdiction. The procedures for obtaining consent will therefore have to be approved for each jurisdiction, and will be described in separate standard operating procedures. It is noted that legal restrictions in some EU Member States prevent performing any trial-specific interventions (e.g. treatment or trial-specific diagnostic procedures without obtaining prior informed consent).

If a patient was unable to give consent at trial entry, but regains capacity to receive information and give consent, he/she will be given information as soon as possible and asked whether he/she is willing to continue his/her participation in the trial. The patient and his/her legal representative will be informed of the right to withdraw from the trial and object to the use of his/her data.

# 7.2 Randomisation procedure and recording of baseline characteristics

Patients will be randomly allocated to tenecteplase or control in a 1:1 ratio. Randomisation will be performed by central computer over the Internet. The investigators will record patient details via a secure web interface before randomisation takes place. Investigators may also contact the Trial Coordinating Centre via the 24-hours help-line.

The randomisation procedure will include a standard minimisation algorithm which will ensure that the treatment groups are balanced for key prognostic factors, such as sex, age, NIHSS score, stroke type (OCSP subgroup), delay to thrombolytic treatment, and use of antiplatelet drugs within the past 24 hours. To avoid predictable alternation of treatment allocation, and thus potential loss of allocation concealment, patients will be allocated with a probability of 0.80 to the

treatment group that would minimise the difference between the groups on the key prognostic factors.

#### 8. Trial treatment

Patients will be randomly allocated to open-label tenecteplase plus best standard care or to best standard care alone

## 8.1 Open-label tenecteplase plus best standard care

The total dose of tenecteplase is 0.25 mg per kg of body weight (maximum 25 mg). The dose shall be given as an intravenous bolus. Patients will be on bed rest in accordance with local routine following administration of tenecteplase.

After infusion, vital signs, neurological signs and blood pressure will be monitored every 15 minutes for two hours, then every 30 minutes for 6 hours, than 60 minutes until 24 hours from the start of treatment. Blood pressure should be maintained at or below 180/105 mmHg during the first 24 hours. Placement of intra-arterial catheters, indwelling bladder catheters, and nasogastric tubes shall be avoided for 24 hours if the patient can be safely managed without them. Venipunctures should be performed and monitored carefully.

#### 8.2 Best standard care alone

Patients randomised to control shall not be given tenecteplase or any other thrombolytic agent.

#### 8.3 Best standard care and other treatments

Both arms will receive best standard care, including intra-arterial interventions for proximal cerebral artery occlusion. <sup>63</sup> If the patient is given tenecteplase, then aspirin or other antiplatelet or anticoagulant drugs shall not be given until 24 hours after termination of infusion and after the control CT brain scan. If the patient was allocated to control, he/she will receive aspirin 300 mg as a loading dose as soon as possible after randomisation. After the first 24 hours the recommended daily dose of aspirin is 75 mg once daily in both the tenecteplase group and the control group. Best standard care during the first week also includes treatments to maintain normal homeostasis (temperature, blood glucose, hydration, nutrition), as well as lipid lowering and blood pressure lowering drugs, in accordance with clinical guidelines. Clinical examinations, including additional CT scans will be performed as clinically indicated.

#### 8.4 Management of serious adverse events related to study treatment

The management of serious adverse events that can be related to treatment with tenecteplase will be guided by specific, detailed standard operating procedures. All patients with neurological deterioration will undergo emergency head CT. In case of a major bleeding (e.g. intracranial haemorrhage), antifibrinolytic agents or transfusion of cryoprecipitate, fresh frozen plasma or platelets may be indicated and should be considered. The investigator should institute any supplementary investigations of serious adverse events based on their clinical judgement of the likely causative factors. This may include seeking further opinion from a specialist in the field of the adverse event.

# 9. Visits and examinations from trial entry till end of follow-up

The duration of the follow-up period is 3 months. During this period, all patients should be treated according to standard clinical guidelines, at the discretion of the clinician. Table 2 gives an overview of all visits and examinations in the trial.

Table 2. Scheme for visits and examinations

| | I | Days | Months | |
|---|---|---|---|---|
| | 1 | 2 | 7 | 3 |
| Clinical visit | X | | X | |
| Routine blood analysis | X | | X | |
| CT + CT angiography (if possible) before randomisation | X | | | |
| CT perfusion, at selected centres | (x) | | | |
| CT + CT angiography (if possible) 24±6 hrs after randomisation | | X | | |
| Centralised follow-up | | | | X |

Day 1 is the day of entry into the trial. \*Day 7 or day of discharge, whichever occurs first.

# 9.1 Visits and examinations during stay in hospital

Clinical visits: These will be performed on day 1 (at baseline) and day 7 (or on the day of discharge, whichever occurs first). NIHSS will be performed at both times. ECG will be performed on day 1. Clinical events will be recorded on day 7 (or on the day of discharge). Outcome assessors will be blinded to the assigned treatment group.

Routine blood analysis will be performed on day 1 (at baseline) and day 7 (or on the day of discharge, whichever occurs first). Tests on day 1 will include: haemoglobin, creatinine, blood glucose, platelets, prothrombin time/INR, aPTT, TT and/or eucarin clotting time if it is suspected that the patient is taking direct thrombin inhibitors or direct factor Xa inhibitors.

Non-contrast CT and CT angiography (if possible): All patients will undergo non-contrast CT and CT angiography (if possible) before randomisation, and again at 24±6 hours after randomisation. CT angiography at 24±6 hours will only be performed in patients with a positive finding on CT angiography before randomisation.

CT perfusion will be performed at selected centres.

# 9.2 Centralised follow-up via telephone or mail at 3 months (90 $\pm$ 7 days)

At 90±7 days, the Trial Coordinating Centre will contact patients (or their carers) via telephone (alternatively, via postal mail), blinded to the treatment that the patients received. We may also need to contact the patients' general practitioners and local hospitals to get information from the patients' medical records. We will record information about clinical events, functional status (mRS), activities of daily living (BI), health-related quality of life (EuroQol), and cognitive status (MMSE, TICS-M).

# 9.3 Long-term follow-up by record linkage with central registries

We will collect data up to three years from trial entry, by using record linkage with data from central registries such as national patient registries and the cause-of-death registries in the participating countries.

#### 10. Effect variables

#### 10.1 Primary effect variable

Functional outcome (defined by the mRS) at 3 months

#### 10.2 Secondary effect variables

#### Clinical events:

- Any intracranial haemorrhage during follow-up
- Symptomatic intracranial haemorrhage by SITS-MOST definition<sup>66</sup>
- Symptomatic intracranial haemorrhage by IST-3 definition<sup>1</sup>
- Parenchymal haemorrhage type 2<sup>67</sup>Stroke progression during follow-up
- Recurrent ischaemic stroke during follow-up
- Major extra cranial bleeding
- Death from all cause during follow-up

Clinical events are defined in the Appendix.

#### Clinical outcomes:

- Favourable functional outcome at 3 months: mRS 0-1
- Good functional outcome at 3 months: mRS 0-2
- NIHSS score at 24 hours and day 7
- Change in NIHSS score from baseline to 24 hours an day 7
- Barthel Index score at 3 months
- EuroOol score at 3 months
- MMSE score at 3 months

#### Radiological outcomes

Radiological outcomes will be defined in a separate imaging protocol.

#### Health-economic variables:

Costs related to:

- Length of hospital stay
- Nursing home care after discharge
- Re-hospitalisations during first 3 months

# 11. Analysis and statistical considerations

#### 11.1 Estimation of sample size

It is uncertain whether the difference in treatment effect between thrombolysed and non-thrombolysed wake-up stroke patients will be similar to that of stroke patients with known time of onset. We originally based our sample size estimation on the results of a Cochrane systematic review of the effect of rt-PA within 4.5 hours of stroke onset, <sup>64</sup> assessed as a binary endpoint (favourable outcome mRS 0-2 versus mRS 3-6). As the primary endpoint in TWIST is mRS across the full ordinal scale (shift analysis), sample size estimation based on ordinal logistic regression analysis is more appropriate.

Longer time from stroke onset to treatment in wake-up stroke patients compared to patients with known symptom onset is anticipated and this is likely to weaken the treatment effect. However, recent trials on patients with wake-up strokes found similar and actually larger differences between thrombolysed and non-thrombolysed patients with wake-up stroke/unknown stroke onset time. In the largest randomized controlled trial on wake-up strokes, WAKE-UP, with favourable outcome defined as mRS 0-1, the difference between thrombolysed and non-thrombolysed patients was 11.5%. The same difference of 11.5% was also found in a recent meta-analysis of 6 observational studies on patients with unknown stroke onset time, where favourable outcome was

defined as mRS 0-2.<sup>65</sup> The MRI-based inclusion criteria in WAKE-UP compared to the CT-based inclusion in TWIST could lead to a smaller treatment effect in TWIST. Furthermore, selection bias in observational studies may result in larger treatment effect than in randomised-controlled trials. It is therefore possible that the effect size in TWIST will be closer to the observed effect in recent studies on wake-up stroke patients than to the effect in previous studies on patients with known time of symptom onset and that the mRS distribution in the control group differs from early trials of IV thrombolytic treatment.

Based on these observations, we assume a treatment effect of 10% absolute difference in a binary endpoint setting (mRS 0-1 versus mRS 2-6) and a distribution between modified Rankin Scale categories similar to that of WAKE-UP with 42% with favourable outcome in the non-thrombolysed group vs 52% in the thrombolysed group, which corresponds to an odds ratio of 1.50. We assume a mRS distribution in the control group in six levels (categories 5 and 6 merged) as 15%, 27%, 23%, 17%, 13%, 5%, (similar to the control group the WAKE-UP trial). With a power of 80%, a two-sided significance level of 5%, and an effect size specified as an odds ratio of 1.50 from an ordinal logistic regression model, the estimated sample size is 600. Based on this, the revised target is to recruit 600 patients, i.e. 300 patients in each arm.

#### 11.2 Statistical analyses

A detailed Statistical Analysis Plan has been drawn up and will be published before breaking the randomisation code. We will analyse the data according to the intention-to-treat principle. Functional outcome will be primarily compared between the study groups by means of ordinal logistic regression, after adjustment for covariates. In a secondary analysis, functional outcome will be dichotomised (mRS score 0-1 vs. 2-6) and analysed by means of logistic regression.

For clinical events we will estimate odds ratios and 95% confidence intervals using logistic regression and estimate hazard ratios and 95% confidence intervals using the Cox proportional hazards model, as appropriate. Interactions will be tested using likelihood ratio tests. The risks of clinical events will be compared using Kaplan-Meyer survival analyses and log-rank tests. All analyses will use 5% two-sided level of significance.

We will perform prespecified subgroup analyses of patients with findings suggestive of penumbra (on CT perfusion), of patients included based on presence or absence of DWI/FLAIR mismatch on MRI, of patients with proximal cerebral artery occlusion, and of patients with different time intervals since awakening, controlling for imbalances in baseline characteristics. Subgroup analyses will be prespecified in the Statistical Analysis Plan. Patients treated with intra-arterial intervention for proximal cerebral artery occlusion will also be analysed separately, and the primary effect variable for this analysis will be cerebral arterial patency before intra-arterial intervention.

Any missing components of the baseline NIHSS will be imputed using a regression-based technique, using age and all other components of the NIHSS. A worst-case approach will be used when handling incomplete dates and times for adverse events. For example, events will be assumed to be treatment emergent unless it is clear even from the partial date/time that this is not the case.

As subgroup analyses are of an exploratory nature, no adjustment for multiple comparisons will be made.

# 12. Trial conduct and practices/procedures

## 12.1 Compliance with regulations and guidelines

The trial will conform to the EU Clinical Trials Directive (2001/20/EC) and national applicable regulatory requirements. EudraCT number: 2014-000096-80. ISRCTN number: 10601890. ClinicalTrials.gov number: NCT03181360.

## 12.2 Data protection

Personal identifiers will not be stored together with clinical information about the patient, but will be stored on a separate, password-protected computer with access only for persons in the Trial Coordinating Centre who are responsible for central follow-up. The code linking personal identifiers with clinical data will be destroyed 15 years after the publication of the primary report, of the trial. The procedures for protection of personal information will be approved by the Research Ethics Committee, and data protection officials at the University Hospital of North Norway.

#### 12.3 Ethical conduct

The trial will be conducted in accordance with the MRC Guidelines for Good Clinical Practice in Clinical Trials, the Council of Europe's Convention on Human rights and Biomedicine (CETS No.: 164), the ICH Harmonized Tripartite Guideline for Good Clinical Practice (CPMP/ICH/135/95) and the Declaration of Helsinki (Edinburgh, October 2000).

We will seek informed consent from all patients, and approval from the ethics committees, according to local or national regulations. All patients will be monitored carefully during treatment and follow-up, and procedures for management of adverse drug reactions, unmasking of the trial treatment, and reporting of serious adverse events are given in the protocol. All events will be evaluated, and the trial will be monitored, audited, and inspected according to applicable regulatory requirements.

#### 12.4 Liability

Patients are indemnified by insurance specific for patients participating in trials of an Investigational Medicinal Product (IMP). Patients are also covered for non-negligent liability by the product indemnity provided by the supplier.

# 12.5 Recording and reporting of serious adverse events

Serious adverse events will be recorded in the case report forms. In case of unexpected serious adverse events, the Trial Coordinating Centre should be notified immediately and within 24 hours at the latest, in accordance with the EC guidance document 2011/C 172/01 ("CT-3"). The report of the SAE must include an assessment of whether there is a reasonable possibility that the IMP caused the event.

Reports of suspected unexpected serious adverse reactions (SUSARs), with all relevant information, will be reported in an expedited manner by the Sponsor, to the competent authority, the ethics committee, and the Data Monitoring Committee, according to the EU Clinical Trials Directive (2001/20/EC) and applicable regulatory requirements. Copies of such reports will be sent to the principal investigators and the Sponsor. (Definitions of serious adverse events and SUSARs: See Appendix).

Serious adverse events that are expected will not be reported in an expedited manner by the Sponsor, for example recurrent ischaemic stroke, intracranial haemorrhage, myocardial infarction, or death. These are events that are expected, and that will be reported as end-points in the case

report forms. Expected adverse reactions listed in Section 4.8 of the Summary of Product Characteristics will also not be reported in an expedited manner.

# 12.6 Event adjudication

A central Event Adjudication Committee will evaluate all events, blinded to treatment allocation.

## 12.7 Monitoring of data quality

The central computer randomisation system will check eligibility for all patients entered in the trial. Data entered over the Internet (at trial entry) and data in case report forms will be checked for validity and internal consistency, to ensure high data quality and completeness, and coherence with the protocol. Centres with poor standards will be contacted and appropriate measures will be taken. During the course of the study the Sponsor will visit all centres at start-up and least once for monitoring purposes, with review of the CRF, comparison with source documents, and observation of the conduct of the trial and adherence to the Protocol. It will be particularly important to check that each patient exists, that a valid consent form is present in the hospital notes, to confirm patient information and adherence to the protocol. There will also be frequent telephone contacts, with the purpose of facilitating the work and fulfilling the objectives of the study.

## 12.8 Handling of protocol violations and protocol amendments

The nature and reasons for the protocol violation shall be recorded in the CRF, in the source documents and in the monitoring visit report. All of this serious non-compliance will be followed up and reported to RA and IEC as per local regulations. In parallel, corrective and/or preventive actions will be undertaken and documented, including any retraining of the investigator and site staff. All patients who have been included in the trial will be followed up, irrespective of whether treatment was discontinued prematurely, or whether the protocol was violated. If treatment discontinuations or protocol violations become frequent the Data Monitoring Committee will consider whether there is a need to increase the number of patients to be included in the trial.

All important changes to the trial will be specified in protocol amendments. Amendments must be approved by the Steering Committee, and the Sponsor has the responsibility to seek approval from the competent authorities the ethics committees. Completed and signed protocol amendments will be circulated to all those who were on the circulation list for the original protocol. Amendments will be listed in chapter 17.

#### 12.9 Monitoring of effectiveness and safety

During the course of the trial the Data Monitoring Committee (DMC) will every 6 months perform an unblinded review of SAEs, in all patients, and in the prespecified subgroups. The DMC will also perform an unblinded interim analysis of the primary efficacy and safety variables (functional outcome and intracranial haemorrhage) when half of the patients have been included. If, in their view, there is credible evidence of harm, or overwhelming evidence of efficacy, the committee will advise the chairman of the Steering Committee. Unless this happens, the Steering Committee will remain ignorant of the interim results.

The DMC will also be responsible for monitoring the overall conduct of the trial, and may formulate recommendations relating to the selection, recruitment, or retention of participants, or their management, or to improving their adherence to protocol-specified regimens, and the procedures for data management and quality control.

The DMC will convene before the start of the trial to agree on the exact terms of reference for the committee, and will meet annually during the course of the trial.

.

# 12.10 Audit and inspection

All source data and all trial data and material will be made directly available for audit and inspection. Source data is all information in original records and certified copies of original records that is necessary for the reconstruction and evaluation of the trial.

#### 12.11 Handling of patient data

All patients will be assigned a unique code number. The patient data will be linked to this number, and the patients' names or other personal identifiers will not be included in the database. The patient database will be kept on a separate, secure computer. The code will be stored on another, secure computer, and will be deleted 15 years after the results of the trial have been published. The trial's procedures for data protection will conform to the Norwegian applicable regulatory requirements, and to the conditions set by the Norwegian Data Inspectorate.

#### 12.12 Handling of the list of treatment codes

The lists of random treatment codes will be produced by the Statistical Centre at the University of Tromsø. Copies of the list will be kept by the person setting up the central randomisation system, and the Trial Statistical Centre. The list will be kept secret for all other people involved in the trial until the closure of the patient database.

## 12.13 Screening logs

Participating centres will be asked to make records of all patients considered for inclusion in the trial (screening logs).

#### 12.14 Financial conduct

Contracts will be agreed between the Sponsor and each of the investigators/institutions. The Coordinating Investigator or other people centrally involved in the trial will not have any financial or other conflicts of interest in connection to the trial. Patients participating in the trial will be reimbursed for their travel expenses.

# 12.15 Publication and data sharing policy

The trial will be published in accordance with the CONSORT guidelines and will be presented by a writing committee on behalf of the investigators. All participating centres and collaborators will be acknowledged in the main publication. The primary results and results of any substudies will be presented at international meetings and in public media.

#### 12.16 User involvement

The Patient Advisory Board consists of representatives from two stroke patient organisations in Norway, with Arne Hagen from Norsk forening for slagrammede, and Anne Heimdal from Hjerneslag. The board will be consulted in all phases of the study.

# 13. Central trial organisation

#### 13.1 Sponsors and funding bodies

The University Hospital of North Norway is the Sponsor of the trial. Address: UNN Tromsø, NO-9038 Tromsø, Norway. Telephone number: +47 77626000. The Director of Research will act as the Sponsor's legal representative.

The trial receives basic funding from the Norwegian Ministry of Health and Care Services (Clinical Therapy Research in the Specialist Health Services Research Programme (KLINBEFORSK)) and the National Association for Public Health. The trial also receives funding from the British Heart Foundation and from the Swiss Heart Foundation. Boehringer-Ingelheim GmbH will reimburse the Sponsor for the costs of tenecteplase.

## 13.2 Trial Coordinating Centre

The Trial Coordinating Centre is based at the Brain and Circulation Research Group at the University Hospital of North Norway and the University of Tromsø.

The Trial Coordinating Centre consists of the following persons: Trial Coordinating Investigator and Head of Brain and Circulation Research Group Ellisiv B. Mathiesen, Trial Manager Melinda B. Roaldsen, Trial Officer and postdoc researcher Agnethe Eltoft, Assistant Trial Manager Mary-Helen Søyland, Trial IT Manager David Perry, Trial Research Nurse Tone Bratteng.

Eivind Berge had a central role in the initiation, planning and implementation of the trial and was Trial Co-coordinating Investigator until his death in February 2020.

#### 13.3 Trial Statistical Centre

Tom Wilsgaard (chair), others.

# 13.4 Executive Committee

Melinda Roaldsen, Agnethe Eltoft, Ellisiv B. Mathiesen.

## 13.5 Imaging Scientific Committee

Agnethe Eltoft, Arnstein Tveiten, representatives from other centres/countries.

#### **13.6 Trial Steering Committee**

Bent Indredavik (Chair), Ellisiv B. Mathiesen, Tom G. Robinson, David Werring, Arnstein Tveiten, Jesper Petersson, Erik Lundström, Hanne Krarup Christensen, Jukka Putaala, Janika Kõrv, Dalius Jatuzis, Gian Marco De Marchis, Stefan Engelter, Tom Wilsgaard.

# 13.7 Data Monitoring Committee

Terje R. Pedersen (Chair), Peter Sandercock, Hans Wedel (statistician).

#### 13.8 Event Adjudication Committee

To be appointed.

#### 14. Time table and end of trial

First patient included: July 2017 Last patient included: September 2021 End of follow-up: December 2021 Presentation of main results: 2022

Follow-up by record linkage with central registries: December 2025

The end of the trial is defined as the last visit of the last patient included.

#### 15. References

- 1. IST-3 Collaborative Group. The benefits and harms of intravenous thrombolysis with recombinant tissue plasminogen activator within 6 h of acute ischaemic stroke (the Third International Stroke Trial [IST-3]): a randomised controlled trial. Lancet 2012;379:2352-63. [Erratum, Lancet 2012;380:730.]
- 2. Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, et al. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014;384:1929-1935.
- 3. Bassetti C, Aldrich M. Night time versus daytime transient ischaemic attack and ischaemic stroke: a prospective study of 110 patients. J Neurol Neurosurg Psychiatry. 1999;67:463-467.
- 4. Moradiya Y, Janjua N. Presentation and outcomes of "wake-up strokes" in a large randomized stroke trial: analysis of data from the International Stroke Trial. J Stroke Cerebrovasc Dis. 2013;22:e286-292.
- 5. Wroe SJ, Sandercock P, Bamford J, Dennis M, Slattery J, Warlow C. Diurnal variation in incidence of stroke: Oxfordshire community stroke project. BMJ. 1992;304:155-157.
- 6. Marsh EE 3rd, Biller J, Adams HP Jr, Marler JR, Hulbert JR, Love BB, et al. Circadian variation in onset of acute ischemic stroke. Arch Neurol. 1990;47:1178-1180.
- 7. Marler JR, Price TR, Clark GL, Muller JE, Robertson T, Mohr JP, et al. Morning increase in onset of ischemic stroke. Stroke. 1989;20:473-476.
- 8. Silva GS, Lima FO, Camargo EC, Smith WS, Singhal AB, Greer DM, et al. Wake-up stroke: clinical and neuroimaging characteristics. Cerebrovasc Dis. 2010;29:336-342.
- 9. Roveri L, La Gioia S, Ghidinelli C, Anzalone N, De Filippis C, Comi G. Wake-up stroke within 3 hours of symptom awareness: imaging and clinical features compared to standard recombinant tissue plasminogen activator treated stroke. J Stroke Cerebrovasc Dis. 2013;22:703-8.
- 10. Fink JN, Kumar S, Horkan C, Linfante I, Selim MH, Caplan LR, et al. The stroke patient who woke up: clinical and radiological features, including diffusion and perfusion MRI. Stroke. 2002;33:988-993.
- 11. Mackey J, Kleindorfer D, Sucharew H, Moomaw CJ, Kissela BM, Alwell K, et al. Population-based study of wake-up strokes. Neurology. 2011;76:1662-1667.
- 12. Serena J, Davalos A, Segura T, Mostacero E, Castillo J. Stroke on awakening: looking for a more rational management. Cerebrovasc Dis. 2003;16:128-133.
- 13. Todo K, Moriwaki H, Saito K, Tanaka M, Oe H, Naritomi H. Early CT findings in unknown-onset and wake-up strokes. Cerebrovasc Dis. 2006;21:367-371.
- 14. Manawadu D, Bodla S, Keep J, Jarosz J, Kalra L. An observational study of thrombolysis outcomes in wake-up ischemic stroke patients. Stroke. 2013;44:427-431.
- 15. Barreto AD, Martin-Schild S, Hallevi H, Morales MM, Abraham AT, Gonzales NR, et al. Thrombolytic therapy for patients who wake-up with stroke. Stroke. 2009;40:827-832.
- 16. Meretoja A, Putaala J, Tatlisumak T, Atula S, Artto V, Curtze S, et al. Off-label thrombolysis is not associated with poor outcome in patients with stroke. Stroke. 2010;41:1450-1458.
- 17. Manawadu D, Bodla S, Jarosz J, Kalra L. Thrombolysis in selected patients with wake up stroke is feasible with similar safety as thrombolysis in 0-4.5 hours. Abstract. International Stroke Conference 2012, New Orleans, USA, January 31-February 03, 2012.
- 18. Kim JT, Park MS, Nam TS, Choi SM, Kim BC, Kim MK, et al. Thrombolysis as a factor associated with favorable outcomes in patients with unclear-onset stroke. Eur J Neurol. 2011;18:988-994.
- 19. Song SS, Copen WA, Yoo AJ, Ford AL, Hsia A, Muzikansky A et al. Expanding Opportunities for Intravenous Alteplase Treatment of Patients With Unwitnessed Acute Stroke Using MRI-based Patient Selection: Imaging Results of the MR WITNESS Multicenter Trial (NCT01282242). Abstract - oral presentation. International Stroke Conference 2016, Los Angeles, USA, February 17-19, 2016.

- 20. Thomalla G, Simonsen CZ, Boutitie F, Andersen G, Berthezene Y, Cheng B, et al. MRI-Guided Thrombolysis for Stroke with Unknown Time of Onset. N Engl J Med. 2018:379:611-622.
- 21. Lindekleiv H, Mathiesen EB, Berge E. Recanalisation therapies for wake-up stroke. The Cochrane Library 2014. <a href="http://onlinelibrary.wiley.com/doi/10.1002/14651858.CD010995/abstract">http://onlinelibrary.wiley.com/doi/10.1002/14651858.CD010995/abstract</a>.
- 22. Michel P, Ntaios G, Reichhart M, Schindler C, Bogousslavsky J, Maeder P, et al. Perfusion-CT guided intravenous thrombolysis in patients with unknown-onset stroke: a randomized, double-blind, placebo-controlled, pilot feasibility trial. Neuroradiology. 2012;54:579-588.
- 23. Ma H, Parsons MW, Christensen S, et al. A multicentre, randomized, double-blinded, placebo-controlled Phase III study to investigate EXtending the time for Thrombolysis in Emergency Neurological Deficits (EXTEND). Int J Stroke. 2012;7:74-80.
- 24. Koga M, Toyoda K, Kimura K, Yamamoto H, Sasaki M, Hamasaki T, et al. THrombolysis for Acute Wake-up and unclear-onset Strokes with alteplase at 0·6 mg/kg (THAWS) Trial. Int J Stroke. 2014;9:1117-1124.
- 25. Wake up Symptomatic Stroke Benefit of Intravenous Clot Busters or Endovascular Intervention (WASSABI). ClinicalTrials.gov Identifier: NCT01455935.
- 26. Dunn CJ, Goa KL. Tenecteplase: a review of its pharmacology and therapeutic efficacy in patients with acute myocardial infarction. Am J Cardiovasc Drugs. 2001;1:51-66.
- Tsikouris JP, Tsikouris AP. A review of available fibrin-specific thrombolytic agents used in acute myocardial infarction. Pharmacotherapy. 2001;21:207-217.
- 28. Haley EC Jr, Lyden PD, Johnston KC, Hemmen TM. A pilot dose-escalation safety study of tenecteplase in acute ischemic stroke. Stroke. 2005;36:607-612.
- 29. Matosevic B, Knoflach M, Werner P, Pechlaner R, Zangerle A, Ruecker M, et al. Fibrinogen degradation coagulopathy and bleeding complications after stroke thrombolysis. Neurology. 2013;80:1216-1224.
- 30. Szabo S, Letsch R, Ehlers R, Walter T, Kazmaier S, Helber U, et al. Absence of paradoxical thrombin activation by fibrin-specific thrombolytics in acute myocardial infarction: comparison of single-bolus tenecteplase and front-loaded alteplase. Thromb Res. 2002;106:113-119.
- 31. Benedict CR, Refino CJ, Keyt BA, Pakala R, Paoni NF, Thomas GR, et al. New variant of human tissue plasminogen activator (TPA) with enhanced efficacy and lower incidence of bleeding compared with recombinant human TPA. Circulation. 1995;92:3032-3040.
- 32. Serebruany VL, Malinin AI, Callahan KP, Binbrek A, Van De Werf F, Alexander JH, et al. Effect of tenecteplase versus alteplase on platelets during the first 3 hours of treatment for acute myocardial infarction: The Assessment of the Safety and Efficacy of a New Thrombolytic Agent (ASSENT-2) platelet substudy. Am Heart J. 2003;145:636-642.
- 33. Keyt BA, Paoni NF, Refino CJ, Berleau L, Nguyen H, Chow A, et al. A faster-acting and more potent form of tissue plasminogen activator. Proc Natl Acad Sci U S A. 1994;91:3670-3674.
- 34. Collen D, Stassen JM, Yasuda T, Refino C, Paoni N, Keyt B, et al. Comparative thrombolytic properties of tissue-type plasminogen activator and of a plasminogen activator inhibitor-1-resistant glycosylation variant, in a combined arterial and venous thrombosis model in the dog. Thromb Haemost. 1994;72:98-104.
- 35. Refino CJ, Paoni NF, Keyt BA, Pater CS, Badillo JM, Wurm FM, et al. A variant of t-PA (T103N, KHRR 296-299 AAAA) that, by bolus, has increased potency and decreased systemic activation of plasminogen. Thromb Haemost. 1993;70:313-319.
- 36. Thomas GR, Thibodeaux H, Errett CJ, Badillo JM, Keyt BA, Refino CJ, et al. A long-half-life and fibrin-specific form of tissue plasminogen activator in rabbit models of embolic stroke and peripheral bleeding. Stroke. 1994;25:2072-2078; discussion 2078-2079.
- 37. Chapman DF, Lyden P, Lapchak PA, Nunez S, Thibodeaux H, Zivin J. Comparison of TNK with wild-type tissue plasminogen activator in a rabbit embolic stroke model. Stroke. 2001;32:748-752.

- 38. Lapchak PA, Araujo DM, Zivin JA. Comparison of tenecteplase with alteplase on clinical rating scores following small clot embolic strokes in rabbits. Exp Neurol. 2004;185:154-159.
- 39. Lapchak PA, Araujo DM. Reducing bleeding complications after thrombolytic therapy for stroke: clinical potential of metalloproteinase inhibitors and spin trap agents. CNS Drugs. 2001;15:819-829.
- 40. Lapchak PA, Araujo DM, Pakola S, Song D, Wei J, Zivin JA. Microplasmin: a novel thrombolytic that improves behavioral outcome after embolic strokes in rabbits. Stroke. 2002;33:2279-2284.
- 41. Lapchak PA, Araujo DM, Song D, Wei J, Zivin JA. Neuroprotective effects of the spin trap agent disodium-[(tert-butylimino)methyl]benzene-1,3-disulfonate N-oxide (generic NXY-059) in a rabbit small clot embolic stroke model: combination studies with the thrombolytic tissue plasminogen activator. Stroke. 2002;33:1411-1415.
- 42. Van de Werf F, Adgey J, Ardissino D, Armstrong PW, Aylward P, Barbash G, et. al. Single-bolus tenecteplase compared with front-loaded alteplase in acute myocardial infarction: the ASSENT-2 double-blind randomised trial. Lancet. 1999;354(9180):716-22.
- 43. Molina C, Ribo M, Rubiera M, Santamarina E, Delgado-Mederos R, Maisterra O. TNK induces faster MCA recanalization and leads to better short- and long-term clinical recanalization and leads to better short- and long-term clinical study [Abstract]. Stroke. 2008;39:563.
- 44. Smadja D, Chausson N, Joux J, Saint-Vil M, Signate A, Edimonana M, et al. A new therapeutic strategy for acute ischemic stroke: sequential combined intravenous tPA-tenecteplase for proximal middle cerebral artery occlusion based on first results in 13 consecutive patients. Stroke. 2011;42:1644-1647.
- 45. Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, et al. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010;41:707-711.
- 46. Parsons MW, Miteff F, Bateman GA, Spratt N, Loiselle A, Attia J, et al. Acute ischemic stroke: imaging-guided tenecteplase treatment in an extended time window. Neurology. 2009;72:915-921.
- 47. Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, et al. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012;366:1099-1107.
- 48. Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, et al. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015;14:368-376.
- 49. Coutts SB, Dubuc V, Mandzia J, Kenney C, Demchuk AM, Smith EE, et al. Tenecteplase-tissue-type plasminogen activator evaluation for minor ischemic stroke with proven occlusion. Stroke. 2015;46:769-774.
- 50. Huang X, Fulton R, Parsons M, et al. Tenecteplase versus Alteplase in acute ischaemic stroke thrombolysis: a meta-analysis of individual patient data from randomised studies. Abstract oral presentation. 1st ESO conference, Glasgow, United Kingdom, April 17-19, 2015.
- 51. Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, et al. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017;16:781-788.
- 52. Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, et al. Tenecteplase versus alteplase before thrombectomy for ischemic Stroke. N Engl J Med. 2018;378:1573-1582.
- Parsons M. Tenecteplase versus Alteplase for Stroke ThrombolysisEvaluation (TASTE) trial. https://www.anzctr.org.au/Trial/Registration/TrialReview.aspx?id=363714.
- 54. A Randomized Controlled Trial of TNK-tPA Versus Standard of Care for Minor Ischemic Stroke With Proven Occlusion (TEMPO-2). ClinicalTrials.gov Identifier: NCT02398656.
- 55. Alteplase-Tenecteplase Trial Evaluation for Stroke Thrombolysis (ATTEST2). ClinicalTrials.gov Identifier: NCT02814409.

- 56. Kidwell CS, Jahan R, Gornbein J, Alger JR, Nenov V, Ajani Z, et al. A trial of imaging selection and endovascular treatment for ischemic stroke. N Engl J Med. 2013;368:914-923.
- 57. Thomalla G, Cheng B, Ebinger M, et al. DWI-FLAIR mismatch for the identification of patients with acute ischaemic stroke within 4·5 h of symptom onset (PRE-FLAIR): a multicentre observational study. Lancet Neurol. 2011;10:978-986.
- 58. Parsons MW, Pepper EM, Bateman GA, Wang Y, Levi CR. Identification of the penumbra and infarct core on hyperacute noncontrast and perfusion CT. Neurology. 2007;68:730-736.
- 59. Hopyan J, Ciarallo A, Dowlatshahi D, Howard P, John V, Yeung R, et al. Certainty of stroke diagnosis: incremental benefit with CT perfusion over noncontrast CT and CT angiography. Radiology. 2010;255:142-153.
- 60. Ezzeddine MA, Lev MH, McDonald CT, Rordorf G, Oliveira-Filho J, Aksoy FG, et al. CT angiography with whole brain perfused blood volume imaging: added clinical value in the assessment of acute stroke. Stroke. 2002;33:959-966.
- 61. Schramm P, Schellinger PD, Klotz E, Kallenberg K, Fiebach JB, Kulkens S, et al. Comparison of perfusion computed tomography and computed tomography angiography source images with perfusion-weighted imaging and diffusion-weighted imaging in patients with acute stroke of less than 6 hours' duration. Stroke. 2004;35:1652-1658.
- 62. Leiva-Salinas C, Wintermark M, Kidwell CS. Neuroimaging of cerebral ischemia and infarction. Neurotherapeutics. 2011;8:19-27.
- 63. Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL.Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418.
- 64. Wardlaw JM, Murray V, Berge E, del Zoppo G, Sandercock P, Lindley RL, et al. Recombinant tissue plasminogen activator for acute ischaemic stroke: an updated systematic review and meta-analysis. Lancet. 2012;379:2364-2372.
- 65. Zhu RL Xu J, Xie CJ, Hu Y, Wang K. Efficacy and safety of thrombolytic therapy for stroke with unknown time of onset: a meta-analysis of observational studies. J Stroke Cerebrovasc Dis. 2020;29:104742
- 66. Wahlgren N, Ahmed N, Davalos A, Ford GA, Grond M, Hacke W, et al. Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet. 2007;369(9558):275-282
- 67. von Kummer R, Broderick JP, Campbell BCV, Demchuk A, Goyal M, Hill MD, et al. The Heidelberg Bleeding Classification: Classification of bleeding events after ischemic stroke and reperfusion therapy. Stroke. 2015; 46:2981–2986.

# 16. Appendix

# 16.1 Completed and on-going studies of thrombolytic treatment for wake-up stroke

| Trial (clinicaltrials.gov ID) | Planned<br>enrolment | Participants | Interventions | Primary outcome | Recruitment period |
|---|---|---|---|---|---|
| WAKE-UP (NCT01525290) | 800 (503<br>enrolled) | Ischaemic<br>stroke;<br><4.5 hours after<br>awakening;<br>MRI<br>DWI/FLAIR<br>mismatch | 1. IV alteplase<br>2. Placebo | mRS score<br>at 90 days | Nov 2012 –<br>June 2017 |
| WASSABI (NCT01455935) | 90 | Ischaemic<br>stroke on wake-<br>up; <24 h of<br>onset; NIHSS 8-<br>22; 18-80 years;<br>Penumbra on<br>CT perfusion | <ol> <li>Best medical care</li> <li>IV alteplase</li> <li>IA treatment</li> </ol> | mRS score<br>at 90 days | Nov 2011 – |
| EXTEND (NCT01580839)* *Not a study of wake-up stroke per se, but 146 (65%) of the included patients had wake-up stroke. | 400, revised<br>target 310 (225<br>enrolled) | NIHSS 4-26;<br>Penumbra<br>mismatch on<br>MRI or CT | IV alteplase Placebo | mRS score<br>at 90 days | June 2010 –<br>June 2018 |
| THAWS (NCT02002325) | 300 (131<br>enrolled) | Initial NIHSS<br>≥5 and ≤25;<br>DWI/FLAIR<br>mismatch on<br>MRI | IV alteplase Control | mRS at 90<br>days | April 2014 –<br>July 2018 |

#### 16.2 Definitions of clinical events

#### 16.2.1 Serious adverse events

A serious adverse event is any untoward medical occurrence that, at any dose:

- results in death
- is life threatening
- requires hospitalisation or prolongation of an existing hospitalization
- results in disability/incapacity
- is a congenital abnormality / birth defect.

Medical and scientific judgement should be exercised in deciding whether reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalisation, but may jeopardise the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These should also be considered serious. Examples of such events are invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation, or development of drug dependency or abuse.

#### 16.2.2 Death

Death will be classified according to cause:

- 1. Initial stroke
- 2. Recurrent stroke
- 3. Myocardial infarction
- 4. Infection
- 5. Other vascular cause (e.g. systemic emboli)

- 6. Other non-vascular cause (e.g. malignancy, trauma)
- 7. Unknown cause

#### 16.2.3 Recurrent stroke

Neurological deterioration (increase of  $\geq 2$  on NIHSS, after exclusion of other causes for neurological deterioration) occurring after 72 hours will be considered as a recurrent stroke. Recurrent stroke will be classified as ischaemic, haemorrhagic or unknown (if not documented on imaging).

#### 16.2.4 Symptomatic intracranial haemorrhage (SICH)

The IST-3¹ and SITS-MOST<sup>66</sup> definition of symptomatic intracranial haemorrhage are used: **SICH per IST-3**: symptomatic intracranial haemorrhage is defined as clinically significant deterioration (neurological deterioration, new headache, new acute hypertension, new nausea or vomiting, or sudden decrease in conscious level) or death within the first seven days of treatment with evidence of either significant brain parenchymal haemorrhage (local or distant from the infarct) or significant haemorrhagic transformation (HT) of an infarct on brain imaging. **SICH per SITS-MOST**: SICH is defined as local or remote parenchymal haematoma type 2 on the imaging scan obtained 22-36 hours after treatment, plus neurological deterioration, as indicated by an increase in National Institutes of Health Stroke Scale (NIHSS) score of ≥4 points compared to baseline value or the lowest value between baseline and 24 (± 6) hours, or haemorrhage leading to death.

**Parenchymal haematoma type 2** indicates a haematoma exceeding 30% of the infarct, with obvious mass effect.67

#### 16.2.5 Asymptomatic intracranial haemorrhage

Intracranial haemorrhage on brain MRI or CT without: neurological deterioration, new headache, new acute hypertension, new nausea or vomiting or sudden decrease in conscious level.

#### 16.2.6 Neurological deterioration due to index stroke

The definition is an increase of  $\geq 2$  points in one or more of the NIHSS (irrespective of improvement in any of the other NIHSS sub-scores). When diagnosing neurological deterioration due to index stroke, systemic reasons for deterioration, such as drug-induced hypotension, drug-induced drowsiness, and intercurrent disease should be excluded. No significant haemorrhage should be found on post randomization CT or MR scan.

#### 16.2.7 Acute myocardial infarction

Either one of the following criteria satisfies the diagnosis of myocardial infarction:

- 1. Typical rise and gradual fall (troponin) or more rapid rise and fall (CK-MB) of biochemical markers of myocardial necrosis with at least one of the following:
  - a. ischaemic coronary symptoms;
  - b. development of pathologic Q waves on the ECG;
  - c. ECG changes indicative of ischemia (ST segment elevation or depression); or
  - d. coronary artery intervention (e. g. coronary angioplasty).
- 2. Autopsy pathologic findings of an acute myocardial infarction.

#### 16.2.8 Major extracranial bleeding

Definition of major extracranial bleeding: Clinically overt bleeding associated with one or more of:

- Transfusion of >2 red cell units of blood
- A decrease in haemoglobin of 20 g/l (=2 g/dl, = 1.24 mmol/l)
- Bleeding into retroperitoneum, intraocular space or major joint
- Bleeding leading to permanent treatment cessation

Otherwise, the bleeding will be characterized as minor.

#### 16.3 Abbreviations

aPTT Activated partial thromboplastin time

ATTEST Alteplase versus tenecteplase for thrombolysis after ischaemic stroke

CONSORT Consolidated Standards of Reporting Trials

CRF Case report form
CT Computed tomography
DWI Diffusion-weighted imaging

ECG Electrocardiography ECT Ecarin clotting time

EXTEND Extending the Time for Thrombolysis in Emergency Neurological Deficits Trial

FLAIR Fluid-attenuated inversion recovery
IEC Independent ethics committee
IMP Investigational medicinal product
INR International normalized ratio
MMSE Mini-mental state examination
MRI Magnetic resonance imaging

MR-RESCUE Mechanical Retrieval and Recanalization of Stroke Clots Using Embolectomy

mRS Modified Rankin Scale

NIHSS National Institutes of Health Stroke Scale NOR-TEST The Norwegian tenecteplase stroke trial

SSS Scandinavian Stroke Scale

TASTE Tenecteplase versus Alteplase for Stroke Thrombolysis Evaluation

THAWS Thrombolysis for Acute Wake-up and Unclear-onset Strokes With Alteplase at

0.6 mg/kg Trial Thrombin time

WAKE-UP Efficacy and Safety of MRI-based thrombolysis in Wake Up Stroke

WASSABI Wake Up Symptomatic Stroke in Acute Brain Ischemia

# 17. Summary of changes

#### 17.1 Protocol version/date 160323

• Addition of signature page

TT

- Addition of section 3.2: Potential benefits and harms of tenecteplase
- Change to section 4.2 (Study questions and objectives)
- Change to section 5.2 (Exclusion criteria):
  - New exclusion criterion: "NIHSS score >25 or NIHSS consciousness score >2, or seizures during stroke onset"
  - o Change to wording of exclusion criterion "High risk of bleeding"
  - o New exclusion criterion: "Contraindications to tenecteplase"
  - Change to wording of exclusion criterion "Childbearing potential, pregnancy, positive pregnancy test, breastfeeding"
- Change to section 6.1 (Patient screening)
- Change to section 7.1 (Patient information and consent/assent)
- Change to section 7.2 (Randomisation procedure and recording of baseline characteristics)
- Change to section 8 (Trial treatment)
- Change to section 9 (Visits and examinations from trial entry till end of follow-up)
- Change to section 11.2 (Statistical analyses)
- Change to section 12.2 (Data protection)
- Change to section 12.5 (Recording and reporting of serious adverse events)
- Change to section 12.7 (Monitoring of data quality)
- Change to section 12.8 (Handling of protocol violations)
- Change to section 12.9 (Monitoring of effectiveness and safety)
- Change to section 12.10 (Audit and inspection)
- Change to section 16.2 (Definitions of clinical events)

• Change to section 17 (Summary of changes)

#### 17.2 Protocol version/date 160421

• Change to section 7.1 (Patient information and consent/assent)

#### 17.3 Protocol version/date 170412

- Change to front page, signature page, sections 13.1 (Sponsor) and 13.2 (The Trial Coordinating Centre): Change of sponsor
- Change to section 12.2 (Data protection) and 12.11 (Handling of data): Change from "Norwegian Data Inspectorate" to "Data Protection Officials"
- Change to section 12.16 (User involvement): Change in text
- Change to section 13.7 (Data Monitoring Committee): New names

#### 17.4 Protocol version/date 180410

- Change to section 5.2 (Exclusion criteria): Reversal of effect of anticoagulant drugs
- Change to section 10.2 (Secondary effect variables): New timing
- Change to 11.2 (Statistical analyses): Specification of secondary analysis
- Change to section 13.1 (Sponsor and Funders), 13.2 (Trial Coordinating Centre), 13.6 (Trial Steering Committee): Update
- Change to section 14 (Time table): Update

#### 17.5 Protocol version/date 180704

- Section 3: Update on results of recently published relevant studies
- Section 5.1: Change to inclusion criterion: "NIHSS score ≥3"
- Sections 5.2, 6.1 and 8.1.3: Removal of exclusion criterion: "Patient will be treated with intraarterial interventions for proximal cerebral artery occlusion"
- Section 10.2: Change to secondary effect variables
- Section 11.2: Pre-specification of secondary analyses
- Section 13.6: Change to Trial Steering Committee

#### 17.6 Protocol version/date 200131

• Section 14: Update of time table

#### 17.7 Protocol version/date 200917

- Section 5.2: Change to exclusion criteria: the words "or adnexanet" was deleted from the exclusion criterion: "Any known defect in coagulation (...)"
- Section 11.1: Revision of sample size estimation with calculation based on ordinal shift analysis (in line with the primary endpoint in TWIST) and on results from recent studies on patients with wake-up stroke
- Section 12.16: Change to User involvement (update of members of Patient Advisory Board)
- Section 13.1: Correction of Sponsor's address
- Section 13.2: Change to Trial Coordinating Centre
- Section 13.4: Change to Executive Committee
- Section 13.5: Change to Imaging Scientific Board
- Section 13.6: Change to Trial Steering Committee
- Section 13.8: Update of Event Adjudication Committee
- Section 14: Change to time table
- Section 15: Update of references
- Section 16.1: Update of table
- Section 16.2: Specifications and additions to definitions of clinical events